CLINICAL TRIAL: NCT05471193
Title: Prediction of Cardiac Instability in Intensive Care
Acronym: PRECAIN
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PRECAIN
Record Dates: First submitted 2022-07-12; First posted 2022-07-22 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Hemodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Instability
  Interventions: Diagnostic Test: Machine Learning Prediction
- No Instability
  Interventions: Diagnostic Test: Machine Learning Prediction

INTERVENTIONS:
Diagnostic Test: Machine Learning Prediction — Machine Learning Prediction

SUMMARY:
A large number of different organ functions are recorded in real time for patients who are monitored in an intensive care unit. On the one hand, the measured values collected in this way are used for continuous monitoring of vital parameters, but they are also evaluated several times a day in order to be able to make decisions regarding further diagnostics and therapy. In the first case, threshold values can be defined, and if these are exceeded or fallen short of, the treatment team is automatically alerted. If these limits are set too liberally, then the alert will only indicate an acute risk to the patient, where extensive pathophysiological changes have already occurred. If the limits are chosen too restrictively, then there are frequent false alarms, since the limits are exceeded in most cases due to natural fluctuation, without this having any pathological value. The consequence is a so-called "alarm fatigue", which in the worst case leads to ignoring correct alarms and thus endangers the patients. By design, all of these readings only show the status quo of a patient. It is the task of the treatment team to predict from the course of these readings whether a threatening situation is developing for the patient.

For daily clinical practice, it would be better if dangerous changes in vital signs could be predicted. In this case, it would be possible to intervene therapeutically not only when a dangerous situation has arisen, but to try to avert this situation through adequate measures by changing the therapy strategy. In such a case, the treatment team would no longer be confronted with emergency alarms, but could counteract an impending deterioration with a long lead time.

The first approaches for detecting a drop in blood pressure, for example, which are based on simple models, are already in clinical use.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients that have been treated at the intensive care units of the Kepler University Hospital, Linz, Austria between 2018-03-01 and 2020-10-31.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As described in the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 3069 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
AUROC for Classification of Instability | 2018-03-01 to 2020-10-31
  AUROC for Classification of Instability

SECONDARY OUTCOMES:
Confusion Matrix | 2018-03-01 to 2020-10-31
  Confusion Matrix Results: true positives, true negatives, false positive, false negatives and values calculated from these results.
Descriptive Statistics This outcome measure will compare the individual feature (e. g. height in cm) in one group vs. the other. Significant difference will be described by p-value. | 2018-03-01 to 2020-10-31
  Descriptive Statistics (age in years, height in cm, weight in kg, gender as male/female, date of death, standard laboratory measurements (e. g. blood gas analysis, full blood count, liver function tests, kidney function tests), ICD 10-codes associated with the patient's admission, Glasgow Coma Scale)
  This outcome measure will compare the individual feature (e. g. height in cm) in one group vs. the other. Significant difference will be described by p-value.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tschoellitsch, MD, Principal Investigator — Kepler University Hospital and Johannes Kepler University, Linz, Austria
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tschoellitsch T, Kaltenleithner S, Maletzky A, Moser P, Seidl P, Bock C, Thumfart S, Giretzlehner M, Hochreiter S, Meier J. Mean arterial pressure is all you need in a machine learning model for mean arterial pressure prediction. Eur J Anaesthesiol. 2025 Dec 1;42(12):1112-1122. doi: 10.1097/EJA.0000000000002238. Epub 2025 Jul 7. PMID 40726206